CLINICAL TRIAL: NCT07197983
Title: Automation of Oocyte and Embryo Vitrification: a Pilot Study
Brief Title: Automation of Oocyte and Embryo Vitrification
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Conceivable Life Sciences (Industry)
Collaborators: CARE Fertility UK (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CP003; 10111748 (Other Grant/Funding Number: UKRI)
Record Dates: First submitted 2025-09-25; First posted 2025-09-30 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Intervention Model Description: A single cohort of patients undergoing IVF/ICSI treatment has their spare eggs and embryos (those not suitable for treatment) divided for parallel assignment to two study arms. Each patient's samples are split, with some assigned to automated vitrification using the PRESERVE-CR system and some assigned to standard manual vitrification. This parallel design using sibling samples allows direct comparison of the two methods while controlling for patient-specific factors.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Automated Vitrification (Experimental): Oocytes/embryos from a particular donor will be randomized to manual or automated vitrification. There will be no randomization at the patient level
  Interventions: Device: Automated Vitrification
- Manual Vitrification (Active Comparator): Oocytes/embryos from a particular donor will be randomized to manual or automated vitrification. There will be no randomization at the patient level
  Interventions: Device: Manual Vitrification

INTERVENTIONS:
Device: Automated Vitrification — The PRESERVE-CR system performs automated vitrification (ultra-rapid freezing) of human oocytes and embryos using robotic manipulation and computer-controlled timing.
  Arms: Automated Vitrification
Device: Manual Vitrification — Control specimens are vitrified by standard vitrification protocol.
  Arms: Manual Vitrification

SUMMARY:
Purpose: This study aims to test whether a new automated system can freeze human eggs and embryos as effectively as the current manual method performed by laboratory staff.

Background: Currently, freezing eggs and embryos during fertility treatments (IVF/ICSI) is done entirely by hand by skilled embryologists. This manual process is time-consuming, requires extensive training, and outcomes can vary between different staff members. Automating this process could help standardize procedures, reduce costs, and potentially make fertility treatments more accessible to patients.

What is Being Tested: The study will compare an automated freezing system (prototype designation PRESERVE-CR) against the standard manual freezing method. The key research question is: Can the automated system preserve eggs and embryos as successfully as experienced embryologists do by hand?

How It Works: Patients undergoing IVF/ICSI treatment at CARE Fertility Manchester who consent to participate will have their surplus eggs and embryos (those not suitable for their treatment) divided into two groups. Some will be frozen using the traditional manual method, and some using the new automated system. Both groups will then be thawed to measure survival rates. Tests do not encompass any reproductive outcomes or the creation of embryos specifically for this research.

Why This Matters: If successful, automated freezing could help reduce the workload on laboratory staff, standardize the freezing process across different clinics, potentially lower treatment costs, and make fertility treatments available to more people who need them. The study only uses oocytes and embryos which are unsuitable for patient treatment and that would otherwise be discarded, ensuring no impact on participants' actual fertility treatment.

ELIGIBILITY:
Inclusion Criteria:

* BMI: Between 20-35 kg/m²
* Ovarian Reserve: Anti-Müllerian Hormone (AMH) ≥1.5 ng/mL

Exclusion Criteria:

* Low ovarian reserve
* Surgical sperm retrieval required

Ages: 18 Years to 38 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 125 (Estimated)
Dates: Start 2025-10-14 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Cryosurvival | Within 14 days of egg retrieval
  The proportion of eggs and embryos that survive the freezing and thawing process when using the PRESERVE-CR automated system compared to manual vitrification (sibling controls).

SECONDARY OUTCOMES:
Procedural Timing | Within 14 days of egg retrieval.
  Time required to complete automated vs manual vitrification procedures
Morphological Quality Assessment | Within 14 days of egg retrieval
  Visual evaluation of egg/embryo structure and appearance post-thaw
Technical Performance Metrics | Within 14 days of egg retrieval.
  Level of autonomy achieved (percentage of procedures completed without operator intervention outside of UI input). Operator assistance (frequency and type of manual interventions, if any). Success rates of specific robotic actions (picking, placing, plunging).

CONTACTS AND LOCATIONS:
Locations (1):
- CARE Fertility, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in an article, after de-identification (text, tables, figures, and appendices).
  Data sharing is subject to ethical, legal, and privacy considerations. We are committed to following established guidelines and best practices for data sharing.
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal, to achieve aims in the approved proposal.
  Proposals may be submitted up to 36 months following article publication. Proposals should be directed to PI@Conceivable.life; to gain access, data requestors will need to sign a data access agreement.